CLINICAL TRIAL: NCT06102590
Title: Oxygen Extraction-guided Transfusion Strategy in Critically Ill Patients. A Randomized Controlled Trial.
Brief Title: Oxygen Extraction-guided Transfusion
Acronym: OXYTRIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Dr, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OXYTRIP
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized RBCT (Experimental): Requires daily assessment of hemoglobin (Hb) levels. Prescription of RCBT is restricted to patients who present Hb ≤ 9.0 g/dL and O2ER ≥ 30%. If O2ER < 30%, transfusion will take place only when Hb falls below 7.0 g/dL. Further O2ER measurements during the day in this group are allowed, and the clinician should not be blinded of the results. To tolerate Hb levels below 7.0 g/dL with O2ER < 30% remains a clinical decision, documented in the CRF. Transfusion with Hb below 6.0 g/dL is mandatory
  Interventions: Other: Individualized red blood cell transfusion strategy
- Control group (Active Comparator): Requires daily assessment of hemoglobin levels. Prescription of RCBT is restricted to patients who present Hb ≤ 7.0 g/dL, despite of O2ER values. Indeed, O2ER calculation takes place at least once daily in this group but does not interfere with clinical decision to prescribe RBCT. A liberal transfusion threshold (i.e. 9.0 g/dL) is still possible in critically ill adults with acute coronary syndromes, as indicated by the European current guidelines
  Interventions: Other: European guidelines red blood cell transfusion strategy

INTERVENTIONS:
Other: Individualized red blood cell transfusion strategy — Prescription of RCBT is restricted to patients who present Hb ≤ 9.0 g/dL and O2ER ≥ 30%.
  Arms: Individualized RBCT
Other: European guidelines red blood cell transfusion strategy — RBCT according to ESICM guidelines
  Arms: Control group

SUMMARY:
In critically ill patients, optimized strategies for red blood cells transfusion (RBCT) are still controversial. Most recent guidelines suggest that clinical practice in ICU setting should follow a restrictive approach to RBCT (i.e., hemoglonim level < 7.0 g/dL).In our previous study, oxygen extraction ratio (O2ER) has shown good performance as a marker to identify the correct timing for RBCT, potentially affecting 90-day mortality in non-bleeding, critically ill patients [11]. Moreover, our data suggested that an individualized strategy for RBCT may reduce the incidence of acute kidney injury (AKI), which is possibly related to a better delivery of oxygen and organ perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Hb levels ≤ 9.0 g/dL (as confirmed through a blood test and/or through blood gas analysis)
* Presence of an arterial line and a central venous line (either jugular or subclavian), with confirmed correct position of the catheter tip at the atrio-caval junction (allowing correct estimation of central venous saturation, ScvO2).

Exclusion Criteria:

* Age < 18 years;
* Pregnancy
* Clinical evidence of acute bleeding
* Diagnosis of haematological malignancy
* Diagnosis of sickle cell disease, or other diseases exposing the patient to chronic RCBTs
* Acquired or congenital disorders of coagulation
* Patients with ongoing AKI of stage 1 or worse and/or known chronic kidney disease (CKD) of stage G3a or worse, defined as glomerular filtration rate below 60 for a minimum of 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | 7-day after study inclusion
  Primary outcome will be the incidence of AKI, according to KDIGO latest definitions

SECONDARY OUTCOMES:
90-day mortality | 90-day after study inclusion
proportion of patients undergoing RBCT, despite adequate/low O2ER | 28 days
  Patients receiving RBCT with O2ER<30%
SOFA score variations | 5 days
  SOFA score at study inclusion-SOFA score at day 5
variations in myocardial-specific troponin | 24 hours after study inclusion
  variations in myocardial-specific troponin
days on vasopressors | 28 days
  number of days on vasopressor therapy
Major Adverse Kidney Events by 90 days (MAKE90) | 90 days
  composite of death, new renal replacement therapy, or persistent renal dysfunction
ICU mortality | through study completion, an average of 180 days
  ICU mortality
In-hospital mortality | through study completion, an average of 180 days
  In-hospital mortality

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Erasme, Brussels, Belgium
- Italy (3):
  - Università di Ferrara, Ferrara, Ferrara
  - Università di Perugia, Perugia, Italy
  - Anestesia e Rianimazione Cardio-Toraco-Vascolare, Siena

IPD SHARING:
Plan to Share IPD: Yes
To be shared under reasonable requests.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Fogagnolo A, Azzolina D, Taccone FS, Pedarzani E, Pasa G, Marianello D, Valpiani G, Marchesini C, Annoni F, Moureau A, Volta CA, Franchi F, Spadaro S. Oxygen extraction-guided transfusion strategy in critically ill patients: study protocol for a randomised, open-labelled, controlled trial. BMJ Open. 2024 Nov 12;14(11):e089910. doi: 10.1136/bmjopen-2024-089910. PMID 39532348